CLINICAL TRIAL: NCT05209854
Title: Evaluation of the Effectiveness of Therapeutic Management in the Care of Chronic Low Back Pain Patients: a Single-center Observational Study.
Brief Title: Evaluation of Therapeutic Management in Chronic Low Back Pain Patients
Acronym: PREDIPAIN
Status: Recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREDIPAIN
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Seventy-eight percent of the population declares being concerned by pain, directly or indirectly. Chronic pain, defined as pain that has lasted for more than three months, affects more than one third of the French population. The national survey of the French Society for the Study and Treatment of Pain (SFETD), conducted in 2009, reveals that the most widespread chronic pain is low back pain (20%).

Pain not only affects the body, but also destroys the person who endures it. A comparative study by Attal et al. carried out on a sample of 1,591 chronic pain sufferers and 1,237 non pain sufferers shows a major impact of pain on the individual's quality of life (SF12), sleep (MOS sleep) and anxiety and depression (HADS).

The 2009 report of the French National Authority for Health (HAS) shows that chronic pain generates a significant societal cost. Low back pain is the leading cause of activity limitation in people aged 45 to 65, and the third leading cause of chronic disability. It is the leading cause of disability in people under 45 years of age, and the leading cause of work stoppage and occupational disease.

The reference tool for assessing pain is currently the Visual Analogue Scale (VAS). However, several factors considerably limit the relevance of an exclusive use of this tool:

* For the patient: the intensity of pain is objectively influenced by many parameters such as the time of day, stress, position, duration of evolution, mechanical or "neuropathic" character, paroxysms, etc. These are all elements that objectively disrupt the evaluation performed by the VAS. When the subjective and emotional dimension is included in these elements, the cloudiness of "true" perception of such a sensation increases even more.
* Difficulties of evaluation for the carer: carers are therefore confronted with a lack of relevance of objective pain evaluation tools, and researchers have to deal with data that are often not very reproducible. A fortiori, the second problem arising from this concerns the difficulty of comparing the effectiveness of different therapeutic strategies. The VAS cannot, for example, take into account the pain dominance in the case of multi-site pain, nor the surface area of the pain zone or even less its typology or topology. This information is however essential to determine the choice of the most appropriate therapeutic strategy.
* The difficulties of evaluation for the health care system: in fact, beyond the therapeutic wandering imposed on certain patients on a "micro" scale, it must be considered that this randomness of evaluation has an impact on the entire health care system. When a decision has to be made to reimburse a particular expensive drug or implantable medical device for pain relief, this reflection has to be extended to the "macro" level. This review thus reveals a threefold need for innovation in pain assessment: for the patient, for the caregiver and for the healthcare system.

DETAILED DESCRIPTION:
To overcome the limitations of the VAS, the PRISMATICS team has developed a triply patented computerized tactile mapping system.

It allows to take into account the objective parameters of pain intensity and surface in a given individual, in a reliable, reproducible and quantitative way.

The Neuro-Mapping Tool: its purpose is to evaluate very precisely the extent of the patient's painful surface at a given moment.

. This prospective study aims to optimize the care pathway and to introduce rationalization and objectivity in the evaluation of therapies proposed to patients.

This study will help us to test the following hypotheses:

* Sociodemographic, psychological, and physiological factors are associated with patient response to the standard care pathway offered to patients with low back pain.
* The different assessment tools are correlated with their evolution.
* The effect of different therapies varies according to patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age at the time the agreement is made.
* Have had low back pain for more than 3 months.
* Have back pain greater than or equal to 2 on the Visual Analog Scale.
* Free patient, without guardianship or tutelage, nor subordination
* No objection from the patient after clear and fair information about the study

Exclusion Criteria:

* Have a life expectancy of less than 12 months (assessed by the physician) at the time of inclusion.
* Persons benefiting from reinforced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, pregnant or breast-feeding women and finally patients in emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from chronic low back pain, consulting at the pain center of Poitiers and/or in consultation in the department of Neurosurgery of Spine - Neurostimulation - Handicap will be included.
Sampling Method: Probability Sample
Enrollment: 613 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogic Scale (0 to 10 points) | 12 months
  Pain scale: 0 (minimum pain) to 10 (maximum pain)
Oswestry Disability Index (0 to 100%) | 12 months
  The questionnaire consists in 10 items ranging from 0 to 5 where 0 indicates high ability to perform the task associated with the item and 5 indicates the inability to perform the task. Items included pain intensity, degree of disability for personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life and travelling.
Quality of Life (0 to 1) | 12 months
  The questionnaire comprises five items including pain intensity, mobility, self-care, daily activities and psychological state (Anxiety or depression).
  Each item consists in a 5 level Likert scale ranging from "I have no problem" to "I am unable to". The maximum score of 1 indicates the best possible quality of life.
Anxiety and Depression Scale (0 to 24) | 12 months
  The questionnaire consists in 14 items each comprising 4 levels and either representing a symptom of anxiety or depression.
  The total score ranges from 0 to 24 for each category (depression or anxiety). A score of 11 or above indicates a definite symptomatology.
Pain Mapping (cm²) | 12 months
  The patient had to draw on the touch screen interface his/her pain in a pre-determined body (in relation with his/her BMI). Before drawing the painful area, the patient chose the red/orange/dark or light blue colour, depending on the pain intensity.
Patient Global Impression of change (0 to 7 "strong impression of change") | 12 months
  Although widely used in chronic pain clinical trials, the validity of PGIC has not been formally evaluated. PGIC is a 7-point scale, assessing patient's perceived improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel ROULAUD, MSc, Study Director — Poitiers University Hospital
Locations (1):
- Poitiers University Hospital, Poitiers, Vienne, France